CLINICAL TRIAL: NCT04810338
Title: Evaluation of the Pronostic Value of Vascular Refilling Rate on Mortality in Chronic Kidney Disease Patients on Dialysis (Stage 5D)
Brief Title: Study Evaluating the Pronostic Value of Vascular Refilling Rate on Mortality in Chronic Kidney Disease Patients on Dialysis
Acronym: REMVAMIR
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0660
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Disease patient on dialysis (stage 5D); Extracorporeal purification; Sodium
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients received conventional dialysis treatment: All patients received conventional dialysis treatment during an observational period of 3 years

SUMMARY:
Aim of this study is to evaluate in a population of chronic kidney disease patients on dialysis (Stage 5D) during an observational period of 3 years:

* the prognostic value of vascular refilling rate on mortality and on the occurrence of i) cardiovascular events and ii) hospitalization number
* the prognostic value of interdialytic weight gain on mortality and on the occurrence of i) cardiovascular events and ii) hospitalization number
* the prognostic value of perdialytic weight loss on mortality and on the occurrence of i) cardiovascular events and ii) hospitalization number.

ELIGIBILITY:
Inclusion criteria:

* Chronic Kidney Disease patient on dialysis (stage 5D) since at least september 2017 (3 months prior to study start date)
* Anuric patient

Exclusion criteria:

- Chronic Kidney Disease patient on dialysis with residual kidney function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients issued from dialysis units (non profit dialysis centers)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Prognostic value of vascular refilling rate on mortality | 2 years after inclusion
  The refilling rate will be assessed by the ratio of relative blood volume
Prognostic value of vascular refilling rate on mortality | 3 years after inclusion
  The refilling rate will be assessed by the ratio of relative blood volume
Prognostic value of vascular refilling rate on mortality | 3 years after inclusion
  The refilling rate will be assessed by the ratio UF max
Prognostic value of vascular refilling rate on mortality | 2 years after inclusion
  The refilling rate will be assessed by the ratio UF max

SECONDARY OUTCOMES:
Prognostic value of interdialytic weight gain | 2 years after inclusion
  Prognostic value of interdialytic weight gain
Prognostic value of interdialytic weight gain | 3 years after inclusion
  Prognostic value of interdialytic weight gain
Prognostic value of perdialytic weight loss | 2 years after inclusion
  Prognostic value of perdialytic weight loss
Prognostic value of perdialytic weight loss | 3 years after inclusion
  Prognostic value of perdialytic weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul CRISTOL, Prof, Study Director — UH MONTPELLIER
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC